CLINICAL TRIAL: NCT04648150
Title: Evaluation of a Millimeter Wave Emission Bracelet -Type Medical Device for Improving Parkinson's Disease Symptoms: Multicenter, Double-blind Randomized Controlled Trial
Brief Title: Evaluation of a Millimeter Wave Emission Bracelet for Improving Parkinson's Disease Symptoms
Acronym: BOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Remedee SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CHH_2020_32
Record Dates: First submitted 2020-11-19; First posted 2020-12-01 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Experimental arm (VERUM): delivery of an active medical device for a period of 2 months. Then delivery of a second active medical device for a period of 4 months.
  Control arm (SHAM): delivery of an inactive medical device for a period of 2 months of use then delivery of an active medical device from M2 to M6 after inclusion.
Who Masked: Participant, Care Provider, Investigator
Masking Description: ratio 1 :1 in each centre on an online randomization module
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VERUM (Experimental): An active wave emission bracelet for a period of 2 months. Then delivery of a second active medical device for a period of 4 months
  Interventions: Device: Evaluation of a millimeter wave emission bracelet for improving Parkinson's disease symptoms
- SHAM (Sham Comparator): An inactive wave emission bracelet for a period of 2 months of use then delivery of an active medical device from M2 to M6 after inclusion.
  Interventions: Device: Evaluation of a millimeter wave emission bracelet for improving Parkinson's disease symptoms

INTERVENTIONS:
Device: Evaluation of a millimeter wave emission bracelet for improving Parkinson's disease symptoms — Evaluation of a millimeter wave emission bracelet -type medical device for improving Parkinson's disease symptoms: multicenter, double-blind randomized controlled trial

SUMMARY:
Idiopathic Parkinson's disease is a common neurodegenerative disease, with a prevalence of around 2% in people over 65 years of age in France.

This pathology affects the dopaminergic pathway but also other systems: cholinergic, noradrenergic and serotoninergic.

The symptoms of Parkinson's disease are motor but also non-motor with sleep, smell, cognitive, psychiatric, digestive, urinary, dysautonomic, painful disorders. The discomfort can be such that invasive and expensive solutions have been developed. Invasive or expensive techniques (deep brain stimulation, lesional microsurgery by gamma knife or ultrasound, duodopa or apokinon pumps) brought significant benefits to patients. Opportunities for clinical improvement using less expensive and lighter devices should be sought.

The Remedee endorphin band device is a device that emits millimeter-band electromagnetic waves on the wrist. The device stimulates subcutaneous nerve endings and activates a physiological response leading to the release of endorphins in the brain. Endorphins are involved in several physiological processes, including pain control.

Mu-opioid receptor (MOR) agonists do not only relieve pain, but have effects related to mesolimbic dopaminergic pathways. Indeed, the opioid and dopaminergic systems are closely linked at the cellular level. Endorphins, through inhibition of the release of the neurotransmitter GABA upon binding to the μ receptor, are also linked to an increase in dopamine.

DETAILED DESCRIPTION:
Intervention 1 Name : VERUM

Description :

Experimental arm (VERUM): delivery of an active medical device for a period of 2 months. Then delivery of a second active medical device for a period of 4 months.

Intervention 2 Name : SHAM

Description:

Control arm (SHAM): delivery of an inactive medical device for a period of 2 months of use then delivery of an active medical device from M2 to M6 after inclusion

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Follow-up for Parkinson's disease for more than 5 years
* Treatment stable for at least 3 months
* Having retained sufficient autonomy to allow participation in the study
* Hoehn and Yahr score in ON DOPA <4

Exclusion Criteria:

* Genetic forms of the disease
* EVA> 7 over the previous week
* Moderate to severe cognitive impairment
* Pathology or condition (other than Parkinson's disease) that can generate motor disorders
* Allergy to metals and / or silicone
* Dermatological pathology on the wrists
* Metal object at one of the wrists (implanted metal material, piercing)
* Presence of a tattoo on one of the wrists
* Wrist circumference <14.5 cm or> 21 cm i.e. wrist incompatible with the MD template
* Inability of the patient to put on and / or wear the template of the medical device
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Fondation Adolphe de Rothschild, Paris
  - Centre Hospitalier de Voiron, Voiron

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VERUM | SHAM
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VERUM | SHAM | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69.5 [63.0 to 74.0] | 66.5 [57.2 to 70.0] | 68.0 [59.8 to 72.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 14 | 14 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Assessment of the Effectiveness of Two Months of Use of the Remedee Endorphin Band Medical Device in Improving Motor Disorders in Patients With Parkinson's Disease
Description: Decrease of 3.25 points or more in the Movement Disorder Society Unified Parkinson Disease Rating Scale III from inclusion.
  The Movement Disorder Society Unified Parkinson Disease Rating Scale III (MDS-UPDRS III score evaluation) will be performed under ON Dopa conditions and blinded from the randomization arm.
  The MDS-UPDRS III varies from 0 to199, a higher score meaning a worse outcome.
Time Frame: two months after inclusion
Measure: Count of Participants; unit: Participants
Arm/Group | VERUM | SHAM
Number analyzed (Participants) | 30 | 30
Participants | 6 | 13

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | VERUM | SHAM
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/50/NCT04648150/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04648150/SAP_001.pdf